CLINICAL TRIAL: NCT07057856
Title: An Analysis of the Relationship Between the Genetic Polymorphisms of Interleukin 12 Receptor Subunit Beta 1 and Crohn's Disease in Chinese Patients
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2025-01-222
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Extract whole genome DNA from peripheral blood
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CD patients: Some CD patients received UST treatment and the first sufficient dose of UST (6mg/kg) was administered intravenously.
  Interventions: Biological: Ustekinumab (UST)
- normal control: no biological agents treatment

INTERVENTIONS:
Biological: Ustekinumab (UST) — The first sufficient dose of UST (6mg/kg) was administered intravenously at weeks 0
  Groups: CD patients

SUMMARY:
From January 2018 to May 2025, diagnosed CD patients and gender- and age-matched normal controls were collected from Department of Gastroenterology, the Second Affiliated Hospital of Wenzhou Medical University. Our study aimed to explore the associations of interleukin 12 receptor subunit beta 1 (IL-12RB1) gene polymorphisms with the risk and clinicopathological characteristics of Crohn's disease (CD), and to analyze the effects of IL-12RB1 gene variations on the clinical response of ustekinumab (UST) treatment in CD patients at week 8.

DETAILED DESCRIPTION:
From January 2018 to May 2025, diagnosed CD patients and gender- and age-matched normal controls were collected from Department of Gastroenterology, the Second Affiliated Hospital of Wenzhou Medical University. Genotypes of IL-12RB1 were examined by multiplex polymerase chain reaction-ligase detection reaction technique. Unconditional logistic regression analysis was employed to analyze the distribution differences of IL-12RB1 gene polymorphisms between CD group and normal control group, as well as their influences on the clinicopathological characteristics and 8-week clinical response to UST treatment of CD patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed CD based on comprehensive clinical, colonoscopy, histopathological, laboratory, and radiographic examination results

Exclusion Criteria:

* rheumatoid arthritis, systemic lupus erythematosus, intestinal tuberculosis, ischemic enteritis, radiation enteritis, tumors, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There was no statistically significant difference in the gender ratio, average age, and proportion of smokers between CD group and normal control group. All study subjects are from the Zhejiang Han population who are not related by blood
Sampling Method: Probability Sample
Enrollment: 866 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Genotypes of IL-12RB1 | Baseline
  multiplex polymerase chain reaction-ligase detection reaction technique

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No